CLINICAL TRIAL: NCT05291702
Title: Multitract PCNL as One Step for Management of Large Renal Stones
Brief Title: Multitract Percutaneous Nephrolithotomy(PCNL) in Large Renal Stones.
Acronym: PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Mahmoud Ali Abbas, Principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Multitract PCNL
Record Dates: First submitted 2022-01-30; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Staghorn Calculi
Keywords: PCNL
MeSH Terms: conditions — Staghorn Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multitract PCNL patients (Other): Assessment of the multitract PCNL procedure in removal of large renal stones using pneumatic or laser lithotripsy.
  Interventions: Procedure: PCNL

INTERVENTIONS:
Procedure: PCNL — Percutaneous nephrolithotomy ( Extraction of the renal stones using the nephroscope/ Ureteroscope )

SUMMARY:
Investigator aimed to analyze the clinical efficacy and safety of multiple tracts PCNL as one step therapy to treat the staghorn stones or multiple calyceal calculi which are inaccessible by single tract

DETAILED DESCRIPTION:
Staghorn calculi are branched stones either partial or complete occupying the pelvis and one or more of the renal caliceal system that is detected by non contrast computrized tomography (NCCT) and plain on kidney, ureter, urinary bladder (KUB). An untreated staghorn calculus over time can damage the kidney and deteriorate its function and /or cause life threatening sepsis.

Total stone clearance is an important goal to eradicate any infective focus, relieve obstruction and preserve the kidney function.

Based on American Urological Association (AUA) guideline, PCNL is the most effective, safest and minimally invasive treatment option compared to open surgery

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients more than 18 years old.
2. Patients with staghorn stone (partial, complete).
3. Patients with multiple calyceal calculi which are inaccessible by single tract.

Exclusion Criteria:

1. Patients under 18 years old.
2. Patients with renal anomalies.
3. Patients with only function kidney.
4. Patients with distal ureteric obstruction.
5. Patients with radiolucent stone.
6. Patients with febrile urinary tract infection.
7. Patients with abnormal coagulopathy state.
8. Patients refused to participate in this study.
9. pregnancy.
10. Musculoskeletal deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | The participants will be followed for one month after the procedure
  Assessment of the instant postoperative stone free rate and after one month from the procedure for all 40 participants using the postoperative non contrast computerized tomography (NCCT )and plain on kidney , ureter, urinary bladder (KUB )

SECONDARY OUTCOMES:
Postoperative complications | From the start of the operation and till one month after the patient discharge.
  Measuring the postoperative complications rates, classification of the severity of the complications will assess the safety of the procedure.
Operative time | Average of three hours
  Measurment of the time from start of the operation till fixation of nephrostomy tube
Postoperative pain | Within 24 hours postoperative and till the patient discharge
  Measurment of the postoperative pain score using the Visual analogue scale(VAS) that is divided into mild(1-3), moderate(4-6) and sever(7-10) according to the severity of the pain.
Hospital stay | Average of six days
  Postoperative hospital stay of the participants till thier discharge

REFERENCES:
- [Background] Romero V, Akpinar H, Assimos DG. Kidney stones: a global picture of prevalence, incidence, and associated risk factors. Rev Urol. 2010 Spring;12(2-3):e86-96. PMID 20811557
- [Background] Turk C, Petrik A, Sarica K, et al. Urolithiassis. European Association of Urolgy. Accessed: August 23,2019.
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Background] Zhu W, Liu Y, Liu L, Lei M, Yuan J, Wan SP, Zeng G. Minimally invasive versus standard percutaneous nephrolithotomy: a meta-analysis. Urolithiasis. 2015 Nov;43(6):563-70. doi: 10.1007/s00240-015-0808-y. Epub 2015 Aug 5. PMID 26242465